CLINICAL TRIAL: NCT00434148
Title: A Randomized, Double-blind Study to Assess the Safety and Efficacy of Different Dose Levels of Pasireotide (SOM230) Subcutaneous (sc) Over a 6 Month Treatment Period in Patients With de Novo, Persistent or Recurrent Cushing's Disease
Brief Title: Safety and Efficacy of Different Dose Levels of Pasireotide in Patients With de Novo, Persistent or Recurrent Cushing's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSOM230B2305; 2006-004111-22 (EudraCT Number)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Cushing's Disease
Keywords: Cushing's Disease; pasireotide; SOM230
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pasireotide 600 ug (Experimental): At randomization, participants received 600 ug subcutaneously (sc) twice daily (bid). Participants continued at this dose until month 6 if their month 3 mean urinary free cortisol (mUFC) was <= 2 x the upper limit of normal (ULN) and the mUFC was below or equal to their baseline mUFC. Participants not meeting the mUFC criteria at month 3 were unblinded and required to increase their dose to 900ug bid on an open label basis. Participants had the option to continue in the extension phase as long as they did not meet any discontinuation criteria or until pasireotide was available commercially in their country.
  Interventions: Drug: Pasireotide
- Pasireotide 900 ug (Experimental): At randomization, participants received 900 ug subcutaneously (sc) twice daily (bid). Participants continued at this dose until month 6 if their month 3 mean urinary free cortisol (mUFC) was <= 2 x the upper limit of normal (ULN) and the mUFC was below or equal to their baseline mUFC. Participants not meeting the mUFC criteria at month 3 were unblinded and required to increase their dose to 1200 ug bid on an open label basis. Participants had the option to continue in the extension phase as long as they did not meet any discontinuation criteria or until pasireotide was available commercially in their country.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide

SUMMARY:
This study will evaluate the safety and efficacy of two different doses of Pasireotide in patients with de novo or recurrent/persistent Cushing's Disease.

ELIGIBILITY:
Inclusion criteria

* 18 years or greater
* Confirmed diagnosis of ACTH-dependent Cushing's disease
* Not considered candidate for pituitary surgery

Exclusion criteria

* History of pituitary irradiation in the last 10 years
* Cushing's syndrome not caused by pituitary tumor
* Patients with active malignant disease (cancer) in the last 5 years
* Women who are pregnant or lactating

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (62):
- United States (10):
  - Stanford University Medical Center Stanford Cancer Center (3), Stanford, California
  - University Chicago Hospital Dept. of Univ of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute The Melanoma Program, Boston, Massachusetts
  - Columbia University Medical Center- New York Presbyterian Columbia University DeptofMed, New York, New York
  - Cleveland Clinic Foundation Dept. of Cleveland Clinic (6), Cleveland, Ohio
  - Oregon Health & Sciences University Dept.ofOregonHealth&SciencesU., Portland, Oregon
  - University of Texas Southwestern Medical Center Clinical-TranslationalRes.Ctr., Dallas, Texas
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(8), Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Swedish Medical Center Dept.ofSeattle Neuroscience(2), Seattle, Washington
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
- Belgium (2):
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
- Brazil (5):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
- China (3):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Denmark (3):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
- Novartis Investigative Site, Helsinki, Finland
- France (9):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Grenoble Cédex 9
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Toulouse
- Germany (4):
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Athens, GR, Greece
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (8):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Porto, Portugal, Portugal
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Fatih / Istanbul

REFERENCES:
- [Derived] Lacroix A, Gu F, Schopohl J, Kandra A, Pedroncelli AM, Jin L, Pivonello R. Pasireotide treatment significantly reduces tumor volume in patients with Cushing's disease: results from a Phase 3 study. Pituitary. 2020 Jun;23(3):203-211. doi: 10.1007/s11102-019-01021-2. PMID 31875276
- [Derived] Yedinak CG, Hopkins S, Williams J, Ibrahim A, Cetas JS, Fleseriu M. Medical Therapy with Pasireotide in Recurrent Cushing's Disease: Experience of Patients Treated for At Least 1 Year at a Single Center. Front Endocrinol (Lausanne). 2017 Feb 27;8:35. doi: 10.3389/fendo.2017.00035. eCollection 2017. PMID 28289402
- [Derived] Schopohl J, Gu F, Rubens R, Van Gaal L, Bertherat J, Ligueros-Saylan M, Trovato A, Hughes G, Salgado LR, Boscaro M, Pivonello R; Pasireotide B2305 Study Group. Pasireotide can induce sustained decreases in urinary cortisol and provide clinical benefit in patients with Cushing's disease: results from an open-ended, open-label extension trial. Pituitary. 2015 Oct;18(5):604-12. doi: 10.1007/s11102-014-0618-1. PMID 25537481
- [Derived] MacKenzie Feder J, Bourdeau I, Vallette S, Beauregard H, Ste-Marie LG, Lacroix A. Pasireotide monotherapy in Cushing's disease: a single-centre experience with 5-year extension of phase III Trial. Pituitary. 2014 Dec;17(6):519-29. doi: 10.1007/s11102-013-0539-4. PMID 24287689
- [Derived] Petersenn S, Newell-Price J, Findling JW, Gu F, Maldonado M, Sen K, Salgado LR, Colao A, Biller BM; Pasireotide B2305 Study Group. High variability in baseline urinary free cortisol values in patients with Cushing's disease. Clin Endocrinol (Oxf). 2014 Feb;80(2):261-9. doi: 10.1111/cen.12259. Epub 2013 Jul 15. PMID 23746264
- [Derived] Colao A, Petersenn S, Newell-Price J, Findling JW, Gu F, Maldonado M, Schoenherr U, Mills D, Salgado LR, Biller BM; Pasireotide B2305 Study Group. A 12-month phase 3 study of pasireotide in Cushing's disease. N Engl J Med. 2012 Mar 8;366(10):914-24. doi: 10.1056/NEJMoa1105743. PMID 22397653
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com//webapp/etrials/searchTrial.do

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment number reflects the participants who were randomized and received at least one dose of drug.
Pre-assignment Details: A total of 165 participants were randomized, but 1 participant from the 600ug group and 2 participants from the 900ug group were not treated. Participants who completed month 12 and did not enter the extension phase were not counted as discontinuations.
Groups:
- Pasireotide 900 ug: At randomization, participants received 600 ug subcutaneously (sc) twice daily (bid). Participants continued at this dose until month 6 if their month 3 mean urinary free cortisol (mUFC) was <= 2 x the upper limit of normal (ULN) and the mUFC was below or equal to their baseline mUFC. Participants not meeting the mUFC criteria at month 3 were unblinded and required to increase their dose to 1200 ug bid on an open label basis. Participants had the option to continue in the extension phase as long as they did not meet any discontinuation criteria or until pasireotode was available commercially in their country.
Period: Overall Study
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Started | 82 ("Started" indicates Full Analysis Set. Patients randomized and treated.) | 80
Completed Month 12 | 39 | 39
Completed m. 12; Did Not Enter Extension | 13 | 7
Completed Month 12; Entered Extension | 26 | 32
Completed | 13 | 7
Not Completed | 69 | 73
Not completed — Adverse Event | 18 | 18
Not completed — Lack of Efficacy | 25 | 28
Not completed — Withdrawal by Subject | 15 | 15
Not completed — Protocol Violation | 4 | 0
Not completed — Administrative problems | 6 | 10
Not completed — Lost to Follow-up | 0 | 1
Not completed — Condition no longer requires study drug | 1 | 0
Not completed — Abnormal test procedure result | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.97) | 39.9 (10.77) | 40.2 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of mUFC (Urinary Free Cortisol) Responders by Randomized Dose Group
Description: A responder in the primary efficacy analysis was a patient with a mUFC≤ULN at Month 6 and whose dose was not increased prior to Month 6.
Time Frame: 6 months
Population: The full analysis set (FAS) was the primary population for efficacy and consisted of all 162 randomized patients who received at least one dose of paseriotide.
Measure: Number (95% Confidence Interval); unit: Responders
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
Responders | 12 [7.0 to 22.3] | 21 [16.6 to 35.9]

2. Secondary Outcome: Change From Baseline in mUFC
Description: Twenty four hour urine samples were collected to obtain mUFC measurements. A negative change from baseline indicates improvement.
Time Frame: baseline, 3 months, 12 months
Population: Only participants from the full analysis set, who had measurements at baseline and the post baseline time point, were included in the analysis for that post baseline time point. The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: nmol/24h
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
nmol/24h
  month 3 (n=61,62) | -375.8 (631.07) | -343.4 (485.48)
  month 12 (n=37,35) | -572.6 (941.44) | -350.7 (380.25)

3. Secondary Outcome: Time to First UFC Response
Description: Time to first UFC response is defined as the number of months from baseline to first attainment of UFC response.
Time Frame: 12 months
Population: Full Analysis Set (FAS): The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
months | 1.0 [0.9 to 2.7] | 1.0 [0.9 to 2.7]

4. Secondary Outcome: Percent Change From Baseline in Serum Cortisol
Description: Blood samlpes were drawn to obtain serum cortisol levels. A negative change from baseline indicates improvement.
Time Frame: baseline, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
Percent change
  month 0.5 (n=77,76) | -4.0 (28.23) | -10.8 (30.57)
  month 1 (n=78,72) | -7.3 (30.13) | -7.7 (32.00)
  month 1.5 (n=75,71) | -5.5 (27.65) | -7.1 (31.34)
  month 2 (n=73,67) | -0.7 (35.81) | -6.4 (29.75)
  month 2.5 (n=70,67) | -3.3 (31.40) | -10.1 (31.23)
  month 3 (n=70,67) | -2.6 (35.79) | -10.2 (25.60)
  month 4 (n=68,61) | -6.9 (31.88) | -10.8 (28.10)
  month 5 (n=62,58) | -4.3 (36.96) | -10.8 (26.50)
  month 6 (n=59,57) | -5.6 (34.28) | -9.3 (31.45)
  month 7 (n=52,53) | -9.8 (34.44) | -5.8 (26.35)
  month 8 (n=50,46) | -10.2 (30.85) | -9.9 (35.79)
  month 9 (n=46,48) | -5.4 (33.49) | -5.8 (31.56)
  month 10 (n=42,47) | -11.2 (30.25) | -9.3 (28.39)
  month 11 (n=41,41) | -8.2 (38.19) | -14.0 (29.63)
  month 12 (n=39,38) | -11.6 (33.75) | -15.2 (21.99)
  month 15 (n=26,26) | -10.5 (30.14) | -12.5 (29.27)
  month 18 (n=26,25) | -7.6 (40.35) | -17.8 (28.39)
  month 21 (n=21,25) | -12.1 (34.23) | -15.5 (34.94)
  month 24 (n=18,22) | -17.9 (43.46) | -18.1 (34.27)
  month 27 (n=16,18) | -9.0 (41.71) | -12.7 (28.53)
  month 30 (n=14,19) | -22.8 (35.43) | -22.7 (32.46)
  month 33 (n=13,15) | -9.5 (44.64) | -25.2 (25.96)
  month 36 (n=10,13) | -12.7 (65.43) | -13.3 (37.84)
  month 39 (n=10,12) | -26.6 (42.89) | -25.9 (33.15)
  month 42 (n=10,12) | -17.8 (39.54) | -18.1 (35.25)
  month 45 (n=10,11) | -12.5 (44.89) | -8.5 (32.55)
  month 48 (n=9,11) | -19.7 (37.88) | -20.1 (39.42)
  month 51 (n=9,9) | -17.6 (34.60) | -24.0 (31.53)
  month 54 (n=9,9) | -25.0 (30.49) | -6.8 (28.07)
  month 57 (n=8,8) | -11.0 (56.61) | -30.8 (22.21)
  month 60 (n=8,8) | -24.5 (31.89) | -18.9 (22.05)
  month 63 (n=6,7) | -28.6 (31.20) | -24.0 (26.41)
  month 66 (n=4,6) | -6.7 (29.29) | -22.5 (36.19)
  month 69 (n=3,5) | -13.4 (42.68) | -33.6 (10.31)
  month 72 (n=3,4) | -4.5 (40.94) | -22.7 (23.57)
  month 75 (n=2,3) | -63.3 (41.13) | -23.2 (25.71)
  month 78 (n=1,1) | 14.5 (NA) — n=1; therefore, SD does not apply. | -53.3 (NA) — n=1; therefore, SD does not apply.

5. Secondary Outcome: Percent Change From Baseline in Mean Adrenocorticotropic Hormone (ACTH)
Description: Blood samples were drawn to obtain ACTH levels. A negative change from baseline indicates improvement.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
percent change
  month 0.5 (n=78,75) | 9.3 (181.17) | -15.9 (30.75)
  month 1 (n=78,71) | -10.0 (37.29) | -19.1 (30.47)
  month 1.5 (n=74,69) | -13.4 (31.64) | -10.5 (38.05)
  month 2 (n=72,66) | -7.7 (40.86) | -13.2 (35.38)
  month 2.5 (n=69,65) | -8.2 (37.32) | -12.0 (47.02)
  month 3 (n=69,66) | -9.2 (40.85) | -16.3 (31.93)
  month 4 (n=66,61) | -7.2 (38.42) | -12.8 (44.06)
  month 5 (n=62,55) | -3.0 (42.50) | -15.0 (38.89)
  month 6 (n=58,55) | -8.4 (43.61) | -17.3 (35.60)
  month 7 (n=52,52) | -11.4 (45.25) | -14.6 (30.88)
  month 8 (n=48,46) | -5.0 (51.75) | -17.0 (36.87)
  month 9 (n=46,47) | -5.3 (55.27) | -18.2 (35.87)
  month 10 (n=42,46) | -10.2 (48.82) | -18.2 (34.18)
  month 11 (n=42,40) | -11.5 (44.52) | -17.4 (39.06)
  month 12 (n=39,39) | -7.4 (53.83) | -26.5 (33.38)
  month 15 (n=26,26) | -14.5 (43.44) | -16.3 (32.01)
  month 18 (n=26,25) | -5.9 (57.56) | -21.2 (32.91)
  month 21 (n=20,23) | -1.5 (51.52) | -17.3 (34.34)
  month 24 (n=18,21) | -10.9 (47.95) | -18.0 (26.53)
  month 27 (n=16,18) | -10.4 (53.33) | -12.5 (39.39)
  month 30 (n=14,18) | -14.7 (56.17) | -20.0 (40.82)
  month 33 (n=13,14) | -9.4 (55.01) | -2.4 (33.07)
  month 36 (n=10,13) | 19.1 (112.26) | 1.2 (35.33)
  month 39 (n=10,12) | -20.9 (48.68) | -5.3 (40.02)
  month 42 (n=10,12) | -6.7 (59.61) | 2.7 (42.35)
  month 45 (n=9,11) | 11.9 (89.59) | 8.1 (50.09)
  month 48 (n=9,9) | -10.8 (65.52) | 11.7 (55.85)
  month 51 (n=9,9) | 0.0 (65.82) | -3.1 (48.21)
  month 54 (n=9,9) | 4.6 (77.49) | 7.3 (52.94)
  month 57 (n=7,7) | 9.6 (59.86) | -5.0 (45.19)
  month 60 (n=8,8) | 9.6 (61.38) | -1.3 (39.01)
  month 63 (n=6,7) | 11.9 (73.78) | 15.4 (50.66)
  month 66 (n=4,6) | 25.3 (75.31) | 18.3 (61.35)
  month 69 (n=3,5) | 38.9 (78.34) | -1.2 (23.98)
  month 72 (n=3,3) | 35.6 (78.48) | 22.0 (46.15)
  month 75 (n=2,3) | -5.0 (77.78) | 23.1 (110.92)
  month 78 (n=1,1) | 50.0 (NA) — n=1; therefore, SD does not apply. | -11.1 (NA) — n=1; therefore, SD does not apply.

6. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Sitting Sytolic Blood Pressure (SBP) and Sitting Diastolic Blood Pressure (DBP)
Description: Sitting blood pressure assessments were performed at every study visit. A negative change from baseline indicates improvement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
mmHg
  Sitting SBP, month 3 (n=70,67) | -7.4 (17.37) | -9.9 (17.01)
  Sitting SBP, month 6 (n=59,57) | -6.8 (19.35) | -11.4 (15.92)
  Sitting SBP, month 12 (n=39,39) | -2.8 (18.40) | -9.4 (14.61)
  Sitting SBP, month 24 (n=18,23) | -11.6 (12.82) | -11.0 (11.58)
  Sitting SBP, month 36 (n=10,13) | -3.0 (17.08) | -11.5 (16.23)
  Sitting SBP, month 48 (n=9,10) | -12.0 (14.15) | -3.6 (14.56)
  Sitting SBP, month 60 (n=7,8) | -12.8 (17.10) | -2.0 (11.83)
  Sitting DBP, month 3 (n=70,67) | -3.3 (11.01) | -4.1 (13.11)
  Sitting DBP , month 6 (n=59,57) | -4.2 (13.54) | -5.0 (11.56)
  Sitting DBP, month 12 (n=39,39) | -2.0 (11.65) | -5.4 (10.86)
  Sitting DBP, month 24 (n=18,23) | -8.1 (11.35) | -6.4 (9.37)
  Sitting DBP, month 36 (n=10,13) | -6.8 (14.17) | -7.3 (8.25)
  Sitting DBP, month 48 (n=9,10) | -11.7 (12.02) | -1.0 (9.30)
  Sitting DBP, month 60 (n=7,8) | -9.1 (9.79) | 0.7 (7.34)

7. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Body Mass Index (BMI)
Description: BMI was determined by using height and weight measurements. A negative change from baseline indicates improvement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48 and month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
kg/m^2
  month 3 (n=70,67) | -1.0 (1.26) | -1.4 (1.29)
  month 6 (n=59,57) | -1.2 (1.64) | -2.1 (1.72)
  month 12 (n=40,39) | -2.1 (2.19) | -2.8 (2.21)
  month 24 (n=18,23) | -3.4 (2.97) | -3.0 (2.67)
  month 36 (n=10,13) | -2.9 (2.47) | -3.3 (3.48)
  month 48 (n=9,10) | -3.1 (2.14) | -2.4 (2.60)
  month 60 (n=8,8) | -2.8 (1.85) | -2.0 (2.20)

8. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Waist Circumference
Description: Waist circumference was measured with a measuring tape correctly positioned. A negative change from baseline indicates improvement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
cm
  month 3 (n=64,66) | -1.0 (10.47) | -2.2 (5.23)
  month 6 (n=53,54) | -1.9 (8.33) | -3.4 (5.39)
  month 12(n=34,35) | -4.4 (9.40) | -5.6 (7.86)
  month 24 ( n=17,22) | -8.7 (9.54) | -5.1 (10.22)
  month 36 (n=9,13) | -7.8 (10.46) | -6.4 (9.97)
  month 48 (n=8,10) | -8.3 (11.59) | -5.1 (10.03)
  month 60 (n=7,8) | -7.3 (12.08) | -4.6 (10.90)

9. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Total Cholesterol and Triglycerides
Description: Blood samples were drawn to obtain total cholesterol and triglycerides' levels. A negative change from baseline indicates improvement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
mmol/L
  Cholesterol, month 3 (n=70,67) | -0.2 (1.06) | -0.3 (1.01)
  Cholesterol, month 6 (n=59,55) | -0.4 (1.24) | -0.4 (0.98)
  Cholesterol, month 12 (n=40,39) | -0.5 (1.29) | -0.6 (1.18)
  Cholesterol, month 24 (n=18,22) | -0.6 (1.39) | -0.3 (0.81)
  Cholesterol, month 36 (n=10,12) | -0.8 (1.24) | -0.1 (0.64)
  Cholesterol, month 48 (n=9,10) | -0.9 (1.63) | -0.4 (0.80)
  Cholesterol, month 60 (n=8,8) | -1.5 (1.57) | -0.4 (1.00)
  Triglycerides, month 3 (n=70,67) | 0.1 (1.07) | 0.1 (1.01)
  Triglycerides, month 6 (n=59,55) | 0 (0.92) | 0.1 (1.00)
  Triglycerides, month 12 (n=40,39) | -0.1 (0.77) | -0.2 (0.69)
  Triglycerides, month 24 (n=18,22) | 0 (1.05) | 0 (0.82)
  Triglycerides, month 36 (n=10,12) | -0.2 (0.99) | 0.3 (1.38)
  Triglycerides, month 48 (n=9,10) | -0.5 (0.94) | 0.4 (1.32)
  Triglycerides, month 60 (n=8,8) | -0.7 (1.01) | 0.2 (1.02)

10. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Beck Depression Inventory (BDI-II) Score
Description: The BDI-II is a 21 item self-report rating inventory measuring characteristic attitudes and symptoms of depression. The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The scores range as follows:
  0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression. A negative change from baseline indicates imrpovement.
Time Frame: baseline, month 3, month 6, month 12, month 18, month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
score on a scale
  month 3 (n=66,65) | -4.6 (8.29) | -1.9 (9.88)
  month 6 (n=56,55) | -4.6 (9.49) | -5.5 (8.81)
  month 12 (n=38,37) | -4.6 (9.19) | -5.2 (9.94)
  month 18 (n=6,6) | -1.3 (5.24) | -7.8 (5.78)
  month 24 (n=0,1) | NA (NA) — No participants had month 24 values. | -12.0 (NA) — n=1; therefore, SD does not apply.

11. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Ferriman-Galway Hirsutism Score
Description: The Ferriman Gallwey scoring system is used to score the degree of excess male pattern body hair. The scorecard of every body location under survey begins from 0 (no excessive terminal hair growth) to 4 (extensive terminal hair growth) and the numbers are added up to a maximum count of 36. A score >= 6 indicates the hirsutism. A negative change from baseline indicates imrpovement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
score on a scale
  month 3 (n=52,50) | -1.3 (3.02) | -1.3 (3.46)
  month 6 (n=44,47) | -0.9 (2.88) | -2.4 (4.70)
  month 12 (n=30,35) | -1.3 (1.99) | -3.5 (4.65)
  month 24 (n=12,22) | -2.8 (2.72) | -4.0 (4.34)
  month 36 (n=7,12) | -3.7 (2.69) | -3.2 (4.09)
  month 48 (n=6,10) | -6.0 (3.85) | -2.5 (2.84)
  month 60 (n=5,8) | -5.0 (3.32) | -2.9 (3.23)

12. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Bone Mineral Density (BMD)
Description: BMD was measured using Lunar or Hologic dual-energy X-ray absorptiometry (DXA) Instruments. Measurements were done in the lumbar vertebrae (L1-L4), proximal femur (total hip) and proximal femur (femur neck). A negative change from baseline indicates imrpovement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
mg/cm^3
  Lumbar vertebrae, month 3 (n=2,2) | 0 (0.02) | 0 (0)
  Lumbar vertebrae, month 6 (n=47,39) | 0 (0.06) | 0 (0.04)
  Lumbar vertebrae, month 12 (n=33,29) | 0 (0.07) | 0 (0.05)
  Lumbar vertebrae, month 24 (n=16,16) | 0 (0.04) | 0 (0.05)
  Lumbar vertebrae, month 36 (n=8,9) | 0 (0.09) | 0.1 (0.12)
  Lumbar vertebrae, month 48 (n=9,8) | 0 (0.12) | 0 (0.05)
  Lumbar vertebrae, month 60 (n=7,6) | 0 (0.14) | 0 (0.08)
  Proximal femur (total hip), month 3 (2,2) | 0 (0.04) | 0 (0.01)
  Proximal femur (total hip), month 6 (n=46,38) | 0 (0.07) | 0 (0.05)
  Proximal femur (total hip), month 12 (n=33,26) | 0 (0.04) | 0 (0.03)
  Proximal femur (total hip), month 24 (n=16,13) | 0 (0.04) | 0 (0.03)
  Proximal femur (total hip), month 36 (n=8,8) | 0 (0.03) | 0 (0.06)
  Proximal femur (total hip), month 48 (n=8,8) | 0 (0.04) | 0 (0.05)
  Proximal femur (total hip), month 60 (n=7,6) | -0.1 (0.14) | 0 (0.06)
  Proximal femur (femur neck), month 3 (n=2,2) | 0 (0) | 0 (0.03)
  Proximal femur (femur neck), month 6 (n=46,38) | 0 (0.03) | 0 (0.05)
  Proximal femur (femur neck), month 12 (n=33,28) | 0 (0.04) | 0 (0.07)
  Proximal femur (femur neck), month 24 (n=16,14) | 0 (0.05) | 0 (0.04)
  Proximal femur (femur neck), month 36 (n=8,8) | 0 (0.02) | 0 (0.04)
  Proximal femur (femur neck), month 48 (n=9,7) | 0 (0.05) | 0 (0.04)
  Proximal femur (femur neck), month 60 (7,6) | 0 (0.10) | 0 (0.05)

13. Secondary Outcome: Mean Change From Baseline in Clinical Signs and Symptoms of Cushing's Disease: Body Composition
Description: Body composition as in percentage of body fat by region was assessed by total body scan. A negative change from baseline indicates improvement.
Time Frame: baseline, month 3, month 6, month 12, month 24, month 36, month 48, month 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of body fat
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
Percentage of body fat
  Month 3 (n=2,2) | 2.9 (1.48) | 0.3 (0.78)
  Month 6 (n=39,32) | -0.4 (3.77) | -0.9 (4.06)
  Month 12 (n=29,22) | -3.0 (4.23) | -1.6 (4.27)
  Month 24 (n=13,14) | -1.9 (3.24) | -1.9 (5.70)
  Month 36 (n=5,8) | -2.0 (4.20) | -1.1 (4.94)
  Month 48 (n=4,7) | -2.0 (5.07) | 0.1 (5.63)
  Month 60 (n=4,6) | -2.8 (4.64) | -0.5 (4.97)

14. Secondary Outcome: Change From Baseline in Tumor Volume
Description: Pituitary magnetic resonance imaging (MRI) was performed to determine tumor volume. A negative change from baseline indicates imrpovement.
Time Frame: baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
cm^3
  month 6 (n=25, 28) | 9.3 (44.02) | -19.0 (36.82)
  month 12 (n=15, 18) | -8.1 (62.17) | -43.8 (49.47)
  month 18 (n=8, 11) | -18.1 (71.62) | -36.0 (65.42)
  month 24 (n=7, 13) | -27.4 (82.68) | -11.5 (66.28)
  month 30 (n=6, 8) | -52.1 (55.20) | -20.9 (77.16)
  month 36 (n=3, 5) | -94.1 (10.15) | -27.6 (78.86)
  month 42 (n=3, 3) | -95.2 (8.40) | 84.0 (282.60)
  month 48 (n=3, 3) | -20.5 (130.90) | 29.2 (164.67)
  month 54 (n=3, 2) | -29.1 (107.40) | 20.3 (170.15)
  month 60 (n=3, 2) | -13.5 (136.97) | 127.6 (321.88)
  month 66 (n= 1, 1) | -100.0 (NA) — n=1; therefore, SD does not apply. | 269.8 (NA) — n=1; therefore, SD does not apply.
  month 72 (n=1, 0) | 45.6 (NA) — n=1; therefore, SD does not apply. | NA (NA) — No participants in this arm had month 72 values.
  month 78 (n=1, 0) | 77.2 (NA) — n=1; therefore, SD does not apply. | NA (NA) — No participants in this arm had month 78 values.

15. Secondary Outcome: Percentage Change From Baseline in Health Related Quality of Life (HRQL) Score
Description: A Cushing's syndrome health related quality of life (HRQL) questionnaire was completed. The Cushing's Syndrome HRQL questionnaire contains 12 sentences with 5 possible answers each. The answers are based on Likert scales, with 5 response categories: Always, Often, Sometimes, Rarely and Never; or Very much, Quite a bit, Somewhat, Very little, and Not at all. The answers to each of the items are rated on a scale of 1 to 5. "1" corresponds to the response category "Always" or "Very much" and "5" corresponds to the category "Never" or "Not at all". The score is the sum of all item responses and can range from 12 to 60 points. The lower the score, the greater the Cushing's Syndrome impacts on HRQoL. A positive change from baseline indicates improvement.
Time Frame: baseline, 3 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in HRQL score
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Number analyzed (Participants) | 82 | 80
Percentage change in HRQL score
  month 3 (n=67,66) | 20.7 (60.26) | 40.1 (135.47)
  month 6 (n= 55,56) | 19.6 (47.78) | 52.2 (169.47)
  month 12 (n=20,20) | 54.9 (95.83) | 111.5 (266.75)

ADVERSE EVENTS:
Groups:
- Pasireotide 600 ug: At randomization, participants received 600 ug subcutaneously (sc) twice daily (bid). Participants continued at this dose until month 6 if their month 3 mean urinary free cortisol (mUFC) was <= 2 x the upper limit of normal (ULN) and the mUFC was below or equal to their baseline mUFC. Participants not meeting the mUFC criteria at month 3 were unblinded and required to increase their dose to 900ug bid on an open label basis. Participants had the option to continue in the extension phase as long as they did not meet any discontinuation criteria or until pasireotode was available commercially in their country.
- Pasireotide 900 ug: At randomization, participants received 900 ug subcutaneously (sc) twice daily (bid). Participants continued at this dose until month 6 if their month 3 mean urinary free cortisol (mUFC) was <= 2 x the upper limit of normal (ULN) and the mUFC was below or equal to their baseline mUFC. Participants not meeting the mUFC criteria at month 3 were unblinded and required to increase their dose to 1200 ug bid on an open label basis. Participants had the option to continue in the extension phase as long as they did not meet any discontinuation criteria or until pasireotode was available commercially in their country.
Arm/Group | Pasireotide 600 ug | Pasireotide 900 ug
Serious Adverse Events (participants affected / at risk) | 23/82 | 25/80
Other Adverse Events (participants affected / at risk) | 78/82 | 79/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 600 ug (N=82) | Pasireotide 900 ug (N=80)
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Tongue movement disturbance (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 1 | 1
Drug ineffective (General disorders) | 1 | 1
Microlithiasis (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 2
Abscess intestinal (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cervicitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 600 ug (N=82) | Pasireotide 900 ug (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 4
Sinus bradycardia (Cardiac disorders) | 8 | 2
Vertigo (Ear and labyrinth disorders) | 4 | 6
Hypothyroidism (Endocrine disorders) | 3 | 4
Vision blurred (Eye disorders) | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 19 | 21
Abdominal pain upper (Gastrointestinal disorders) | 11 | 8
Constipation (Gastrointestinal disorders) | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 49 | 46
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Faeces soft (Gastrointestinal disorders) | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 40 | 47
Vomiting (Gastrointestinal disorders) | 3 | 9
Asthenia (General disorders) | 13 | 6
Fatigue (General disorders) | 12 | 24
Injection site haemorrhage (General disorders) | 1 | 4
Injection site pain (General disorders) | 3 | 4
Malaise (General disorders) | 2 | 5
Oedema peripheral (General disorders) | 9 | 6
Cholelithiasis (Hepatobiliary disorders) | 25 | 25
Gastroenteritis (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 10 | 5
Nasopharyngitis (Infections and infestations) | 12 | 12
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Urinary tract infection (Infections and infestations) | 4 | 6
Contusion (Injury, poisoning and procedural complications) | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 4
Alanine aminotransferase increased (Investigations) | 12 | 6
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 6 | 1
Blood glucose increased (Investigations) | 6 | 3
Blood insulin decreased (Investigations) | 1 | 4
Electrocardiogram QT prolonged (Investigations) | 5 | 7
Gamma-glutamyltransferase increased (Investigations) | 11 | 7
Glycosylated haemoglobin increased (Investigations) | 10 | 8
International normalised ratio increased (Investigations) | 1 | 4
Lipase increased (Investigations) | 7 | 5
Low density lipoprotein increased (Investigations) | 5 | 3
Prothrombin time prolonged (Investigations) | 2 | 4
Weight decreased (Investigations) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 8 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 17 | 18
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 35
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 6
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 10 | 5
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4
Dizziness (Nervous system disorders) | 9 | 9
Dysgeusia (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 25 | 25
Migraine (Nervous system disorders) | 0 | 4
Somnolence (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 6 | 10
Depression (Psychiatric disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 3
Hypertension (Vascular disorders) | 10 | 8
Hypotension (Vascular disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.